CLINICAL TRIAL: NCT03417037
Title: A Phase 3 Open Label, Randomized Study of BMS-986205 Combined With Nivolumab With or Without Chemotherapy Versus Chemotherapy in Participants With Previously Untreated Stage IV or Recurrent Non-Small Cell Lung Cancer
Brief Title: An Immuno-Therapy Study of Experimental Medication BMS-986205 Given With Nivolumab With or Without Chemotherapy Compared to Chemotherapy in Participants With Previously Untreated Stage IV or Recurrent Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA017-062; 2017-003058-18 (EudraCT Number)
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — linrodostat; Nivolumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): BMS-986205 and Nivolumab administered in combination
  Interventions: Drug: BMS-986205; Biological: Nivolumab
- Arm B (Experimental): BMS-986205 and Nivolumab administered in combination with chemotherapy
  Interventions: Drug: BMS-986205; Biological: Nivolumab; Drug: Chemotherapy
- Arm C (Active Comparator): Chemotherapy administered alone
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: BMS-986205 — Administered orally daily, 100 mg
  Arms: Arm A; Arm B
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Arm A; Arm B
Drug: Chemotherapy — Platinum-based doublet chemotherapy
  Arms: Arm B; Arm C

SUMMARY:
This is a study of experimental medication BMS-986205 given with Nivolumab with or without chemotherapy compared to chemotherapy in participants with previously untreated stage IV or recurrent non-small cell lung cancer.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically confirmed stage IV NSCLC per the 8th IASLC of squamous or nonsquamous histology
* Locally advanced disease with recurrence after chemoradiation therapy (stage IIIB disease, specifically refers to patients with no curative treatment options)
* No prior systemic anti-cancer therapy (including EGFR and ALK/ROS1 inhibitors) given as primary therapy for advanced or metastatic disease
* Participants must have biomarker test results available for randomization
* ECOG Performance Status of ≤ 1
* Measurable disease by CT or MRI per RECIST 1.1 criteria

Exclusion Criteria:

* Participants with known sensitizing EGFR mutations or known ALK/ROS1 rearrangements
* Participants with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Participants with an active, known or suspected autoimmune disease [Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll]
* Participants with untreated CNS metastases are excluded [Participants are eligible if CNS metastases are adequately treated and participants are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to first treatment]

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-24 (Estimated); Primary Completion 2021-04-25 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) measured by number of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) divided by the number of randomized participants for each treatment group | 24 months
Progression free survival (PFS) measured by the time between the date of randomization and the first date of documented progression, as determined by the Blinded Independent Central Review, or death, due to any cause, whichever occurs first | 34 months

SECONDARY OUTCOMES:
Overall survival (OS) measured by the time between the date of randomization and the date of death due to any cause | Approximately 5 years
Number of treatment-related adverse events (AE) | Approximately 5 years
Number of treatment-related serious adverse events | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (80):
- United States (19):
  - Local Institution, San Diego, California
  - Local Institution, Fort Myers, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, St. Petersburg, Florida
  - Local Institution, Tallahassee, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution, Decatur, Georgia
  - Local Institution, Marietta, Georgia
  - Local Institution, Wichita, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Boston, Massachusetts
  - Local Institution, Bridgeton, Missouri
  - Local Institution, Lincoln, Nebraska
  - Local Institution, Cleveland, Ohio
  - Local Institution, Gettysburg, Pennsylvania
  - Local Institution, Greenville, South Carolina
  - Local Institution, Lebanon, Tennessee
  - Local Institution, Fort Worth, Texas
  - Local Institution, Lubbock, Texas
- Australia (5):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Melbourne, Victoria
  - Local Institution, Murdoch, Western Australia
  - Local Institution, North Tamworth
- Austria (2):
  - Local Institution, Vienna
  - Local Institution, Wels
- Brazil (8):
  - Local Institution, Ipatinga, Minas Gerais
  - Local Institution, Jd. Petropolis-Londrina, Paraná
  - Local Institution, Centro-porto Alegre, Rio Grande do Sul
  - Local Institution, Ijuí, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Barretos, São Paulo
  - Local Institution, Morumbi, São Paulo
  - Local Institution, Rio de Janeiro
- Local Institution, Québec, Quebec, Canada
- Local Institution, Prague, Czechia
- France (8):
  - Local Institution, Besançon
  - Local Institution, La Tronche
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Pringy
  - Local Institution, Rennes
  - Local Institution, Saint-Herblain
  - Local Institution, Toulon
- Germany (10):
  - Local Institution, Berlin
  - Local Institution, Gauting
  - Local Institution, Gera
  - Local Institution, Göttingen
  - Local Institution, Großhansdorf
  - Local Institution, Hamburg
  - Local Institution, Heidelberg
  - Local Institution, Oldenburg
  - Local Institution, Paderborn
  - Local Institution, Wiesbaden
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Thessaloniki
- Italy (6):
  - Local Institution, Modena
  - Local Institution, Monza (MB)
  - Local Institution, Napoli
  - Local Institution, Perugia
  - Local Institution, Ravenna
  - Local Institution, Reggio Emilia
- Japan (4):
  - Local Institution, Fukushima, Fukushima
  - Local Institution, Morioka, Iwate
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution, Kitaadachi-gun, Saitama
- Local Institution, Mérida, Yucatán, Mexico
- Local Institution, Seoul, South Korea
- Spain (6):
  - Local Institution, A Coruña, Galicia
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Majadahonda - Madrid
  - Local Institution, Málaga
  - Local Institution, Valencia
- Local Institution, Basel, Switzerland
- Local Institution, Taipei, Taiwan
- Turkey (Türkiye) (4):
  - Local Institution, ?stanbul
  - Local Institution, Adana
  - Local Institution, Antalya
  - Local Institution, Istanbul

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx